CLINICAL TRIAL: NCT06670989
Title: Training to Modify Fixational Eye Movements for Optimizing Visual Performance
Brief Title: Training to Modify Fixational Eye Movements for Optimizing Visual Performance in People With Central Vision Loss
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Susana Chung, Professor, National Eye Institute (NEI)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: R21EY030253 (NIH)
Record Dates: First submitted 2024-10-29; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Central Vision Loss From Macular Diseases
Keywords: fixational eye movements; microsaccades; saccade adaptation; fixation training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microsaccade adaptation (Experimental): A fixation target will be presented at the center of the display and participants will be asked to keep the target visible at all time. The investigators will measure participants' fixational eye movements continuously and when a microsaccade (small fast eye movements that occur during fixation of a visual target) is detected, the fixation target (a small dot) will jump to a different location, depending on whether the training is to adapt the microsaccades to have smaller or larger amplitudes. With trials, participants would automatically correct for the spatial errors and thus adapting their microsaccade amplitudes. Training consists of 5-6 sessions of training (about 1 hour each). These training sessions will be scheduled weekly if possible, but it is alright if the sessions are not exactly weekly.
  Interventions: Behavioral: Fixation training

INTERVENTIONS:
Behavioral: Fixation training — Training (adapting) microsaccades during fixation

SUMMARY:
People with central vision loss almost all have exaggerated fixational eye movements when compared with people with normal vision (e.g. larger amplitudes of microsaccades and ocular drifts). Central vision loss primarily results from eye diseases or disorders that affect the macular region of the retina, such as age-related macular degeneration (AMD) and Stargardt disease. The clinical wisdom is that exaggerated fixational eye movements are detrimental to vision. This forms the basis of the increasing number of clinical trials that use fixation stability (variability of eye positions during fixation) as an outcome measure to evaluate the effectiveness of interventions on age-related macular degeneration or other retinal diseases, despite the lack of causal evidence supporting or refuting a relationship between fixational eye movements and functional vision. If excessive fixational eye movements are indeed detrimental to vision for people with central vision loss, can we reduce the amount of their fixational eye movements, thus improve their fixation stability? And if so, does that lead to improved functional vision? The goal of this study is to examine the hypothesis that retinal image motion due to abnormal fixational eye movements can be modified through fixation training, with accompanied improvements in functional vision as a result.

ELIGIBILITY:
Inclusion Criteria:

Participants with normal vision:

* age 18 or above
* best corrected visual acuity of at least 20/20 in each eye
* cataracts, if present, must be minimal (grade 1 or below according to the Lens Opacity Classification System)
* normal contrast sensitivity for their ages
* stereoacuity at least 40 seconds of arc
* no history or signs of any retinal diseases

Participants with macular disorders:

* age 18 or above
* macular disorder present in both eyes
* presence of at least one scotoma within the central 5 degrees of the visual field and with best corrected visual acuity of at least 20/400 in the better-seeing eye
* no foveal island of vision left (i.e. absolute scotoma must include the foveal area)
* cataracts, if present, must be grade 2 or lower according to the Lens Opacity Classification System II

Exclusion Criteria:

Participants with normal vision:

* younger than 18 years of age
* best corrected visual acuity worse than 20/20 in each eye
* cataracts worse than grade 1 according to the Lens Opacity Classification System II
* abnormal contrast sensitivity for their ages
* stereoacuity worse than 40 seconds of arc
* history or signs of any retinal diseases

Participants with macular disorders:

* younger than 18 years of age
* macular disorder absent in at least one eye
* no scotoma within the central 5 degrees of the visual field in the better-seeing eye
* best corrected visual acuity of worse than 20/400 in the better-seeing eye
* foveal island of vision
* cataracts worse than grade 2 according to the Lens Opacity Classification System II

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fixation stability | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Eye positions measured while participants looked at a stationary fixation target for 10 seconds, quantified as the area that captures 68% of eye positions (unit: deg^2).

SECONDARY OUTCOMES:
Visual acuity | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Smallest letter that can be read on an acuity chart (Bailey-Lovie acuity chart). Unit of measurement will be in the logarithm of the minimum angle of resolution (logMAR).
Contrast sensitivity | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  The faintest (lowest contrast) letter that can be read using the Mars Contrast Sensitivity Test. Unit of measurement will be in the logarithm of the contrast sensitivity ("log units").
Reading performance: Maximum reading speed | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Maximum reading speed (unit: words per minute) measured using the MNREAD Acuity Chart (MNREAD Acuity Chart is the name of the instrument that will be used).
Reading performance: critical print size | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  The smallest print size (unit: logMAR) on the MNREAD Acuity Chart that still allow participants to read at their maximum reading speed.
Orientation judgement accuracy: low spatial-frequency | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Accuracy for judging the orientation (tilted to the left or right) of a low spatial-frequency grating. Unit of measurement will be in proportion-correct.
Orientation judgement accuracy: high spatial-frequency | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Accuracy for judging the orientation (tilted to the left or right) of a high spatial-frequency grating. Unit of measurement will be in proportion-correct.
Characteristics of fixational eye movements: microsaccade rate | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Fixational eye movements during the 10 seconds when participants are asked to fixate a target for fixation stability measurement (primary measurement) will be analyzed. The rate of microsaccades (fast eye movements during fixation) will be measured (unit: number per second).
Characteristics of fixational eye movements: microsaccade amplitude | Data will be collected immediately before (within 1 hour) the first training session and immediately after (within 1 hour) the last training session. Data will be reported when analysis is completed for all participants (target date: by June 2025).
  Fixational eye movements during the 10 seconds when participants are asked to fixate a target for fixation stability measurement (primary measurement) will be analyzed. The amplitude of microsaccades (fast eye movements during fixation) will be measured (unit: degrees).

CONTACTS AND LOCATIONS:
Locations (1):
- Herbert Wertheim School of Optometry & Vision Science, University of California Berkeley, Berkeley, California, United States

IPD SHARING:
Plan to Share IPD: No
We will report summary results for the group. Some of the outcome measures are health related and we would like to protect the participants' privacy.